CLINICAL TRIAL: NCT04418999
Title: Safety and Efficacy of Intracanalicular Dexamethasone Insert Compared to Loteprednol Etabonate Ophthalmic Gel 0.38% in Patients With Keratoconus Wearing Gas Permeable Contact Lenses Who Have Been Diagnosed With Allergic Conjunctivitis
Brief Title: Safety and Efficacy of Intracanalicular Dexamethasone Compared to Loteprednol Etabonate in Patients With Keratoconus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Illinois College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19027
Record Dates: First submitted 2020-05-27; First posted 2020-06-05 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2022-08

CONDITIONS: Keratoconus; Dry Eye; Allergy
MeSH Terms: conditions — Keratoconus; Dry Eye Syndromes; Hypersensitivity | interventions — Calcium Dobesilate; Loteprednol Etabonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone insert (Experimental): Per participant, one eye will be randomized to receive the intracanalicular dexamethasone insert at the baseline visit (study eye). DEXTENZA is an ophthalmic insert that is inserted in the lower lacrimal punctum into the canaliculus at the day 1 visit by pulling the lower lid taught and using a forceps to insert the medication into the lower canaliculus through the lower punctum.
  Interventions: Drug: dexamethasone ophthalmic insert 0.4 mg, for intracanalicular use
- Loteprednol etabonate ophthalmic gel 0.38% (Active Comparator): Per participant, one eye will be randomized to receive the standard of care topical lotemax etabonate ophthalmic gel 0.38% (control eye). Patients will be prescribed a loteprednol etabonate ophthalmic gel 0.38% and will instill one drop into the eye following a 4x/day,3x/day,2x/day,1/xday weekly taper
  Interventions: Drug: Loteprednol Etabonate 0.38% Ophthalmic Gel/Jelly

INTERVENTIONS:
Drug: dexamethasone ophthalmic insert 0.4 mg, for intracanalicular use — Experimental
  Other Names: Dextenza
  Arms: Dexamethasone insert
Drug: Loteprednol Etabonate 0.38% Ophthalmic Gel/Jelly — Active Comparator
  Other Names: Lotemax
  Arms: Loteprednol etabonate ophthalmic gel 0.38%

SUMMARY:
Drug delivery platforms are an innovative exciting advancement in ophthalmology. They allow patients to eliminate topical medications which are generally associated with lack of compliance, difficulty of use and requiring help from family members. These delivery systems can be applied easily in office, and patients do not have to worry about drop insertion in their post-operative regimen.

The results of this research project should help to answer the following question: Does the use of a physician administered intracanalicular dexamethasone insert improve the signs and symptoms of ocular allergy and dry eye disease in KC patients compared to the use of topical loteprednol etabonate ophthalmic gel 0.38%?

DETAILED DESCRIPTION:
This prospective, open-label, single-center, randomized, fellow-eye, investigator-sponsored clinical study seeks to investigate the safety and efficacy of the dexamethasone insert in the treatment of allergic conjunctivitis and DED signs and symptoms in patients with Keratoconus using RGP contact lenses when compared to topical standard of care loteprednol etabonate ophthalmic gel 0.38%.

Patients with keratoconus who present for their routine visit who have signs and symptoms of dry eye and allergies, will be asked if they want to participate in the study. After screening a given patient for inclusion and exclusion criteria, and gaining informed consent, one eye will be randomized to receive the dexamethasone insert as determined by a coin flip at the screening visit. The remaining eye will be prescribed a loteprednol etabonate ophthalmic gel 0.38% following a 4,3,2,1 weekly taper. Per enrolled eye, the study period will last for approximately 90 days, consisting of five visits. At Screening/ Baseline, Day 0, Day 7, Day 30 and Day 90, primary and secondary endpoints will be assessed alongside standard-of-care procedures. Adjusting for enrollment period, the study will last a total of approximately 3 months

Inclusion Criteria

A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* 18 years of age or older
* Bilateral Keratoconus
* Bilateral RGP contact lenses
* Bilateral allergic conjunctivitis as determined by the Papillae Efron Scale score of at least 1 and symptoms of itching
* Bilateral underlying dry eye disease as determined by the NEI Fluorescein Staining Scale score of at least 1 and a TBUT of less than 10 and must correlate with dryness on OSDI

Exclusion Criteria

A patient who meets any of the following criteria will be excluded from the study:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Obstructed nasolacrimal duct in the study eye(s)
* Hypersensitivity to dexamethasone
* Patients being treated with immunomodulating agents in the study eye(s)
* Patients being treated with immunosuppressants and/or oral steroids Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Study Procedures Screening/Baseline (Visit 1)

After the patient has provided informed consent, the following information will be collected:

* Inclusion/Exclusion
* Demographics
* Medical History and Concurrent Illnesses
* Concomitant Medications
* Uncorrected and best-corrected visual acuity with manifest refraction as measured by ETDRS chart at 4 meters
* Ophthalmic Examination (with or without dilation)
* QOL assessment as measured by OSDI questionnaire
* Osmolarity (Needs to be done prior to any drop instillation)
* MMP9 (Needs to be done prior to any drop instillation)
* Grading of itching (scale 0-4)
* Papillae conjunctivitis assessment (Efron Scale)
* Conjunctival Injection
* Corneal Staining
* TBUT
* Intraocular Pressure

Insertion Visit/Day 0 (Visit 2)

* Concomitant Medications
* Uncorrected and best-corrected visual acuity with manifest refraction as measured by ETDRS chart at 4 meters
* Ophthalmic Examination (with or without dilation)
* QOL assessment as measured by OSDI questionnaire
* Osmolarity (Needs to be done prior to any drop instillation)
* MMP9 (Needs to be done prior to any drop instillation)
* Grading of itching (scale 0-4)
* Papillae conjunctivitis assessment (Efron Scale)
* Conjunctival Injection
* Corneal Staining
* TBUT
* Intraocular Pressure
* Insertion of Dextenza (intracanalicular dexamethasone insert)
* Insert Visualization
* Subject reported AEs after insertion
* Physician ease of insertion grading

Day 7 (Visit 3)

* Concomitant Medications
* Uncorrected and best-corrected visual acuity with manifest refraction as measured by ETDRS chart at 4 meters
* Ophthalmic Examination (with or without dilation)
* QOL assessment as measured by OSDI questionnaire
* Osmolarity (Needs to be done prior to any drop instillation)
* MMP9 (Needs to be done prior to any drop instillation)
* Grading of itching (scale 0-4)
* Papillae conjunctivitis assessment (Efron Scale)
* Conjunctival Injection
* Corneal Staining
* TBUT
* Intraocular Pressure
* Insert Visualization
* Subject reported AEs after insertion

Day 30 (Visit 4)

* Concomitant Medications
* Uncorrected and best-corrected visual acuity with manifest refraction as measured by ETDRS chart at 4 meters
* Ophthalmic Examination (with or without dilation)
* QOL assessment as measured by OSDI questionnaire
* Osmolarity (Needs to be done prior to any drop instillation)
* MMP9 (Needs to be done prior to any drop instillation)
* Grading of itching (scale 0-4)
* Papillae conjunctivitis assessment (Efron Scale)
* Conjunctival Injection
* Corneal Staining
* TBUT
* Intraocular Pressure
* Insert Visualization
* Subject reported AEs after insertion

Day 90 (Visit 5) or Early Termination

* Concomitant Medications
* Uncorrected and best-corrected visual acuity with manifest refraction as measured by ETDRS chart at 4 meters
* Ophthalmic Examination (with or without dilation)
* QOL assessment as measured by OSDI questionnaire
* Osmolarity (Needs to be done prior to any drop instillation)
* MMP9 (Needs to be done prior to any drop instillation)
* Grading of itching (scale 0-4)
* Papillae conjunctivitis assessment (Efron Scale)
* Conjunctival Injection
* Corneal Staining
* TBUT
* Intraocular Pressure
* Insert Visualization
* Subject reported AEs after insertion
* COMTOL

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Bilateral Keratoconus
* Bilateral RGP contact lenses
* Bilateral allergic conjunctivitis as determined by the Papillae Efron Scale score of at least 1 and symptoms of itching
* Bilateral underlying dry eye disease as determined by the NEI Fluorescein Staining Scale score of at least 1 and a TBUT of less than 10 and must correlate with dryness on OSDI

Exclusion Criteria:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Obstructed nasolacrimal duct in the study eye(s)
* Hypersensitivity to dexamethasone
* Patients being treated with immunomodulating agents in the study eye(s)
* Patients being treated with immunosuppressants and/or oral steroids Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Harthan, Principal Investigator — Illinois College of Optometry
Locations (1):
- Illinois Eye Institute, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 36 eyes completed
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Dexamethasone Insert | Loteprednol Etabonate Ophthalmic Gel 0.38%
Started | 18; 18 Eyes | 18; 18 Eyes
Completed | 18; 18 Eyes | 18; 18 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: 18 participants total one eye received dexamethasone insert; one eye received loteprednol etabonate ophthalmic gel
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Insert | Loteprednol Etabonate Ophthalmic Gel 0.38% | Total
Number analyzed (Participants) | 18 | 18 | 18
Number analyzed (eyes) | 18 | 18 | 36
Age, Categorical [Count of Units; unit: eyes]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 4 | 4 | 8
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 18
Count of eyes [Count of Units; unit: eyes] | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Determine the Effect of Dexamethasone Intracanalicular Insert on Patients With Keratoconus Who Also Have Allergies
Description: For patients with keratoconus who wear contact lenses and suffer with allergies Ocular Surface Disease Index (OSDI) questionnaire will be taken, grading of hyperemia, papillary reaction, corneal staining, and intraocular pressures (IOP) will be taken at each visit The primary outcome measure is papillary grade. This is measured on a grading scale of 0-4. Grade 0 is the lowest score, meaning no papillae are present. Grade 4 is the worse score.
  Papillary grade scale = 0-4 (grade 4 is worse score)
Time Frame: 90 days
Population: 18 eyes per arm/group analyzed (36 eyes total/18 participants total)
Measure: Mean (Standard Deviation); unit: papillary grade
Units Other Than Participants: eyes
Arm/Group | Dexamethasone Insert | Loteprednol Etabonate Ophthalmic Gel 0.38%
Number analyzed (Participants) | 18 | 18
Number analyzed (eyes) | 18 | 18
papillary grade | 1.67 (0.67) | 2 (0.76)

2. Primary Outcome: Determine the Effect of Dexamethasone Intracanalicular Insert on Patients With Keratoconus Who Also Have Elevated Osmolarity
Description: For patients with keratoconus who wear contact lenses and suffer with allergies OSDI questionnaire will be taken, grading of hyperemia, papillary reaction, corneal staining, and IOP will be taken at each visit.
  This outcome is measuring Osmolarity which is measured on a scale in units of milliosmoles. The scale measured is between 250-400 with the higher number being the worse score.
Time Frame: 90 days
Population: 18 eyes per arm/group
Measure: Mean (Standard Deviation); unit: milliosmoles
Units Other Than Participants: eyes
Arm/Group | Dexamethasone Insert | Loteprednol Etabonate Ophthalmic Gel 0.38%
Number analyzed (Participants) | 18 | 18
Number analyzed (eyes) | 18 | 18
milliosmoles | 297.8 (31.6) | 304.5 (21.6)

3. Primary Outcome: Determine the Effect of Dexamethasone Intracanalicular Insert on Patients With Keratoconus and Intraocular Pressure
Description: For patients with keratoconus who wear contact lenses and suffer with allergies OSDI questionnaire will be taken, grading of hyperemia, papillary reaction, corneal staining, and IOP will be taken at each visit.
  This specific measure is measuring intraocular pressure by method of Goldman applanation tonometry. This is measured as a unit measure in units of mmHg between 10-22mmHg.
Time Frame: 90 days
Population: 18 eyes per arm/group
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Dexamethasone Insert | Loteprednol Etabonate Ophthalmic Gel 0.38%
Number analyzed (Participants) | 18 | 18
Number analyzed (eyes) | 18 | 18
mmHg | 14.7 (3.1) | 15.1 (3.1)

4. Primary Outcome: Determine the Effect of Dexamethasone Intracanalicular Insert on Patients With Keratoconus and Dry Eye
Description: For patients with keratoconus who wear contact lenses and suffer with allergies OSDI questionnaire will be taken, grading of hyperemia, papillary reaction, corneal staining, and IOP will be taken at each visit.
  tear-break-up time is measured on a scale of 0-4, the higher the number, the worse the score corneal staining is measured on a scale of 0-4, the higher the number the worse the score
Time Frame: 90 days
Population: 18 eyes per arm/group
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Dexamethasone Insert | Loteprednol Etabonate Ophthalmic Gel 0.38%
Number analyzed (Participants) | 18 | 18
Number analyzed (eyes) | 18 | 18
score on a scale
  Tear Break-Up-Time (scale 0-4) | 3.4 (1.7) | 3.6 (1.8)
  Corneal Staining (Scale 0-4) | 5.0 (2.2) | 5.2 (2.1)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Dexamethasone Insert | Loteprednol Etabonate Ophthalmic Gel 0.38%
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04418999/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT04418999/ICF_001.pdf